CLINICAL TRIAL: NCT00328835
Title: Optic Nerve Compliance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Vision Research Trust (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: ONCS
Record Dates: First submitted 2006-05-18; First posted 2006-05-22 (Estimated); Last update posted 2006-10-17 (Estimated); Status verified 2006-05

CONDITIONS: Glaucoma
Keywords: Optic Nerve; Glaucoma
MeSH Terms: conditions — Glaucoma

INTERVENTIONS:
Procedure: Brief Elevation of IOP

SUMMARY:
Chronic glaucoma is one of the leading causes of blindness and visual loss in the developed world. It is a condition where long term exposure to high eye pressures (intra-ocular pressure) damages the nerve fibres in the eye. This damage can be seen by examiners as changes in the optic nerve. The exact mechanism of how the high intra-ocular pressure causes nerve damage is unknown. Both physiological and mechanical mechanisms are thought to play a role. Previous authors have reported structural changes in the connective tissue of optic nerves of eyes with glaucoma. Structural changes in the optic nerve head which affect the mechanical compliance of the nerve may be significant in the cause of glaucomatous nerve damage. This study aims to assess the compliance of the optic disc in subjects with and without glaucoma. We would test compliance by imaging the optic discs of participants before and during a brief (less than two minutes) increase in intra-ocular pressure. We would aim to repeat the tests on the same subjects 3 years later to see how compliance changed. We would also seek to correlate other important parameters such as corneal thickness and visual field changes with our findings

DETAILED DESCRIPTION:
Chronic glaucoma is one of the leading causes of blindness and visual loss in the developed world (the following reference gives rate of visual impairment/blindness caused by glaucoma in one cross-section of an older Australian population as 6% - Foran S, Wang JJ, Mitchell P. Causes of visual impairment in two older population cross-sections: the Blue Mountains Eye Study. Ophthalmic Epidemiol. 2003 Oct;10(4):215-25). Glaucoma is a condition where long term exposure to high eye pressures (intra-ocular pressure) damages the nerve fibres in the eye. The exact mechanism of how the high intra-ocular pressure causes nerve damage is unknown (Albon J, Purslow PP, Karwatowski WS, Easty DL. Age related compliance of the lamina cribrosa in human eyes. Br J Ophthalmol. 2000 Mar;84(3):318-23). Both physiological and mechanical mechanisms are thought to play a role. Previous authors have reported structural changes in the connective tissue of optic discs of eyes with glaucoma, and postulated that this may contribute to changes in the compliance of the optic nerve head (Pena JD, Netland PA, Vidal I, Dorr DA, Rasky A, Hernandez MR. Elastosis of the lamina cribrosa in glaucomatous optic neuropathy. Exp Eye Res. 1998 Nov;67(5):517-24). Structural changes in the optic nerve head which affect the mechanical compliance of the nerve may be significant in the cause of glaucomatous nerve damage. This study aims to assess the compliance of the optic disc in subjects with and without glaucoma. We would test compliance by imaging the optic discs of participants before and during a brief increase in intra-ocular pressure. We would aim to repeat the tests on the same subjects 3 years later to see how the optic nerve compliance changed. We would also look to correlate changes with other ocular parameters such as corneal thickness and visual field defects.

1. Non-glaucoma group

   Inclusion criteria:

   Age over 18

   Exclusion criteria:

   Previous eye surgery Best corrected visual acuity <6/9 Chronic eye disease (including glaucoma) Glaucomatous optic disc Ocular perfusion abnormalities (e.g. previous retinal artery or vein occlusion; or abnormal vasculature including those whose retinal circulation might be compromised by pressure on the eye).
2. Glaucoma group

Inclusion criteria:

Age over 18 Diagnosis of glaucoma (visual field proven) Stable, well controlled glaucoma

Exclusion criteria:

Secondary glaucoma (eg uveitis, neovascular glaucoma, etc) Advanced or fixation-threatening visual field changes Previous eye surgery Chronic eye disease (not including glaucoma) Ocular perfusion abnormalities (e.g. previous retinal artery or vein occlusion; or abnormal vasculature including those whose retinal circulation might be compromised by pressure on the eye).

Two different groups of participants will be studied, those with glaucoma, and those without glaucoma. Participants will have a routine eye examination performed by an experienced doctor. Information such as visual acuity, intra-ocular pressure, corneal thickness, and optic nerve appearance will be obtained. Then participants will have their optic nerves imaged by a Heidelberg retinal tomograph (HRT). The intra-ocular pressure will then be artificially raised to approximately 50 mmHg for approximately two to four minutes using a suction cup oculopressor. The optic nerve will be imaged again by the HRT during that time. From the HRT images we will calculate the optic nerve compliance using measures such as mean position of the disc, and optic cup area and volume. This data will then be analysed statistically to look for a significant difference in the optic nerve compliance of the two groups. Participants will then undergo the same testing procedure 3 years later to see how their optic nerve compliance has changed. We will then examine these changes to see how they correlate with changes in their vision. These changes would include: development of glaucoma; decreased visual acuity; reduced visual field.

Clinical methods - history and examination. Visual field testing (in those with glaucoma) using an automated visual field testing machine.

Intra-ocular pressure measurement using a Goldmann tonometer. Corneal thickness measurement using a "Pachmate", pachymeter. Optic disc images using a Heidelberg retinal tomograph (a confocal scanning diode laser ophthalmoscope).

There is a theoretical risk that a short term rise in intra-ocular can compromise the blood supply to the optic nerve and cause optic nerve damage. However a previous study looking at optic nerve compliance found no side-effects after a short term rise in intraocular pressure induced with a suction cup (Augusto, A., Harris, A., Cantor, L., Abreu, M., & Weinland, M. Effects of short term increase of intraocular pressure on optic disc cupping. British Journal of Ophthalmology. 1998. 82, 880-883). Also a recent study has shown that a short term rise in intra-ocular pressure does not alter the response of retinal and optic nerve head blood flow (Garhofer, G., Resch, H., Weigert., Lung, S., Simader, C. & Schmetterer, L. Short-term increase of intraocular pressure does not alter the response of retinal and optic nerve head blood flow to flicker stimulation. Investigative Ophthalmology & Visual Science. 2005. 46(5), 880-883). We also know from clinical experience that patients with short term rises in intra-ocular pressure caused by vitreo-retinal surgery and acute angle closure glaucoma do not have long term side effects from raised pressure for hours.

To further reduce the risk of side-effects we will exclude those with advanced or fixation threatening glaucoma changes. We will also exclude those whose retinal circulation is seen to be compromised by digital pressure on the eye during examination.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18, Diagnosis of glaucoma (visual field proven), Stable, well controlled glaucoma

Exclusion Criteria:

* Previous eye surgery, Best corrected visual acuity <6/9, Chronic eye disease (including glaucoma, Secondary glaucoma (eg uveitis, neovascular glaucoma, etc), Advanced or fixation-threatening visual field changes, Ocular perfusion abnormalities (e.g. previous retinal artery or vein occlusion; or abnormal vasculature including those whose retinal circulation might be compromised by pressure on the eye).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-03; Study Completion 2006-04

PRIMARY OUTCOMES:
Optic Disc Change
Visual Field Progression

SECONDARY OUTCOMES:
Visual Acuity Change

CONTACTS AND LOCATIONS:
Overall Officials: Anthony P Wells, FRANZCO, Principal Investigator — CVRT, Wellington School Of Medicine - University of Otago
Locations (1):
- Capital Vision Research Trust, Wellington, New Zealand

REFERENCES:
- [Derived] Poostchi A, Wong T, Chan KC, Kedzlie L, Sachdev N, Nicholas S, Garway-Heath DF, Wells AP. Optic disc diameter increases during acute elevations of intraocular pressure. Invest Ophthalmol Vis Sci. 2010 May;51(5):2313-6. doi: 10.1167/iovs.09-3756. Epub 2009 Nov 11. PMID 19907027
- [Derived] Wells AP, Garway-Heath DF, Poostchi A, Wong T, Chan KC, Sachdev N. Corneal hysteresis but not corneal thickness correlates with optic nerve surface compliance in glaucoma patients. Invest Ophthalmol Vis Sci. 2008 Aug;49(8):3262-8. doi: 10.1167/iovs.07-1556. Epub 2008 Mar 3. PMID 18316697